CLINICAL TRIAL: NCT01366924
Title: The Effect of Amino Acid Supplementation on Skeletal Muscle Protein Turnover Following Endurance Exercise
Brief Title: Essential Amino Acids Supplementation and Muscle Protein Synthesis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: Tufts University (Other)
Responsible Party: Stefan M Pasiakos/Research Physiologist, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H06-04; 7906 Tufts
Record Dates: First submitted 2011-06-01; First posted 2011-06-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2011-06

CONDITIONS: Muscle Loss; Muscle Anabolism
Keywords: protein turnover; whole body protein turnover; essential amino acids; leucine
MeSH Terms: conditions — Muscular Atrophy | interventions — Amino Acids, Essential

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Muscle protein turnover and intracellular signaling at rest (No Intervention): Muscle protein turnover and intracellular signaling are measured at rest for comparison to post-exercise muscle metabolism.
- Muscle metabolism after endurance exercise (Active Comparator): Post-exercise muscle protein metabolism was measured to determine if endurance exercise affects muscle metabolism compared to rest.
  Interventions: Dietary Supplement: Essential Amino Acids; Other: Endurance exercise
- Muscle Metabolism after endurance exercise (Experimental): Muscle metabolism response to endurance exercise with essential amino acid supplementation
  Interventions: Dietary Supplement: Essential Amino Acids
- Muscle anabolism after endurance exercise (Experimental): Muscle anabolism after endurance exercise with essential amino acid supplementation.
  Interventions: Dietary Supplement: Essential Amino Acids

INTERVENTIONS:
Dietary Supplement: Essential Amino Acids — 10 Gram Essential Amino Acid solutions with different leucine contents consumed during two identical endurance exercise trials
  Arms: Muscle Metabolism after endurance exercise; Muscle anabolism after endurance exercise; Muscle metabolism after endurance exercise
Other: Endurance exercise — 60 minute endurance exercise session
  Arms: Muscle metabolism after endurance exercise

SUMMARY:
The modern warfighter faces numerous physiological challenges including sleep deprivation, sustained intense physical activity, and caloric restriction, the combined effects of which may result in the loss of lean body mass and decreased physical performance. Dietary interventions may help preserve lean body mass and facilitate recovery from periods of intense physical demand. For example, dietary strategies that increase amino acid availability have been shown to stimulate protein synthesis in skeletal muscle following resistance exercise. Because military tasks also incorporate endurance exercise components, studies regarding the effects of increasing dietary amino acids following endurance exercise are warranted. The objectives of this study are to characterize the effect of endurance exercise on protein synthesis and breakdown as well as the ability of an essential amino acid supplement to influence skeletal muscle protein metabolism and its cellular and molecular regulation following endurance exercise.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 - 35 years
* Weight stable
* Recreationally active with VO2max of 40 - 50 ml/kg/min
* Refrain from taking any NSAIDS or any aspirin-containing medications
* Supervisor approval if a federal employee

Exclusion Criteria:

* Disease or medication that affects macronutrient metabolism and/or the ability to participate in strenuous exercise
* Allergies to foods or medications (including, but not limited to, lidocaine or phenylalanine) to be utilized in the study
* Abnormal PT/PTT test or problems with blood clotting
* Present condition of alcoholism or other substance abuse that compromises exercise capacity
* Musculoskeletal injuries that compromise the ability to exercise
* Pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in muscle protein synthesis after exercise or exercise with amino acid supplementation. | An average change over a 210 minute recovery period from a 60 minute endurance exercise session

SECONDARY OUTCOMES:
Change in intracellular signaling after exercise or exercise with amino acid supplementation. | At 30 minutes and 210 minutes after a 60 minute endurance exercise session

CONTACTS AND LOCATIONS:
Overall Officials: Stefan M Pasiakos, Ph.D., Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (2):
- United States (2):
  - Tufts University, Boston, Massachusetts
  - US Army Research Institute of Environmental Medicine, Natick, Massachusetts

REFERENCES:
- [Background] Pasiakos SM, McClung HL, McClung JP, Margolis LM, Andersen NE, Cloutier GJ, Pikosky MA, Rood JC, Fielding RA, Young AJ. Leucine-enriched essential amino acid supplementation during moderate steady state exercise enhances postexercise muscle protein synthesis. Am J Clin Nutr. 2011 Sep;94(3):809-18. doi: 10.3945/ajcn.111.017061. Epub 2011 Jul 20. PMID 21775557
- [Result] Pasiakos SM, McClung HL, McClung JP, Urso ML, Pikosky MA, Cloutier GJ, Fielding RA, Young AJ. Molecular responses to moderate endurance exercise in skeletal muscle. Int J Sport Nutr Exerc Metab. 2010 Aug;20(4):282-90. doi: 10.1123/ijsnem.20.4.282. PMID 20739716
- [Result] Scofield DE, McClung HL, McClung JP, Kraemer WJ, Rarick KR, Pierce JR, Cloutier GJ, Fielding RA, Matheny RW Jr, Young AJ, Nindl BC. A novel, noninvasive transdermal fluid sampling methodology: IGF-I measurement following exercise. Am J Physiol Regul Integr Comp Physiol. 2011 Jun;300(6):R1326-32. doi: 10.1152/ajpregu.00313.2010. Epub 2011 Mar 9. PMID 21389329